CLINICAL TRIAL: NCT00084032
Title: A Randomized, Multicenter Trial to Determine Whether Induction Therapy Followed by Treatment Interruption is Superior to Induction Therapy Alone in the Treatment of Primary HIV Infection (PHI): The Structured Treatment Interruption (STI) Study
Brief Title: Anti-HIV Medications and Structured Treatment Interruptions for People Recently Infected With HIV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIEDRP AIN502
Record Dates: First submitted 2004-06-04; First posted 2004-06-07 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Interruption; Treatment Naive; Primary HIV Infection; PHI
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

ARMS (2):
- 1 (Experimental): In Step 1, participants will receive ARV therapy for 24 weeks. Upon entering Step 2, participants will continue taking ARV therapy for 16 weeks and then stop ARVs for 64 weeks.
  Interventions: Behavioral: Structured treatment interruption; Drug: Antiretroviral regimen
- 2 (Experimental): In Step 1, participants will receive ARV therapy for 24 weeks. Upon entering Step 2, participants will stop ARVs for 4 weeks, take ARVs for 8 weeks, stop ARVs for 4 weeks, take ARVs for 8 weeks, and then stop ARVs for 56 weeks.
  Interventions: Behavioral: Structured treatment interruption; Drug: Antiretroviral regimen

INTERVENTIONS:
Behavioral: Structured treatment interruption — Treatment interruption schedule is dependent on the Arm in which participants are enrolled in Step 2
Drug: Antiretroviral regimen — Participants will take any combination of FDA-approved ARV medications prescribed by their physician

SUMMARY:
People recently infected with HIV who are treated with anti-HIV medications may develop strong immune system responses to HIV and may be able to control the virus without continuing to take these medications. The purpose of this study is to see if giving anti-HIV medications to people soon after they have been infected with HIV can help them control HIV. The study will also see if the immune system can control the amount of HIV virus in the blood (viral load) even after a person has stopped taking the medications. The study will evaluate three different schedules of stopping and starting anti-HIV medications to see which schedule is best able to boost a patient's immune system to control HIV viral load.

Hypothesis: Combination therapy started in primary HIV infection, in conjunction with structured treatment interruptions, will result in greater control of viremia off treatment than induction therapy alone.

DETAILED DESCRIPTION:
Initiation of treatment during acute HIV infection seems to result in greater suppression of viral replication than noted during chronic infection and better recovery of certain CD4 subpopulations. However, it is difficult for patients treated during acute infection to maintain long-term continuous antiretroviral (ARV) treatment because of difficulty adhering to complicated medication regimens, drug-related toxicities, and cost of medications. Acutely infected patients who have undergone early initiation of treatment followed by structured treatment interruptions (STIs) appear to have lower off-treatment viral loads than historical controls. This study will evaluate whether effective ARV treatment during acute and early HIV infection followed by STI will result in lower viral setpoints than would otherwise be expected.

This trial will have 2 steps and will last for a maximum of 104 weeks. Participants will either enter Step 1 and continue on to Step 2 or enter Step 2 directly. During Step 1, participants with acute or early HIV infection will be given 24 weeks of ARV therapy. Participants may take any combination of FDA-approved ARV medications that they and their doctors select. Participants will have study visits at study entry and Weeks 1, 4, 8, and 20. After 24 weeks on Step 1, participants may enroll in Step 2.

Participants in Step 1 and people with early or acute HIV infection who began ARV treatment within 21 days of diagnosis and have had no more than 1 year of treatment may enroll in Step 2. During Step 2, participants will be randomly assigned to one of two study arms:

* Arm 1: Participants will continue taking ARV therapy for 16 weeks and then stop ARVs for 64 weeks.
* Arm 2: Participants will stop ARVs for 4 weeks, take ARVs for 8 weeks, stop ARVs for 4 weeks, take ARVs for 8 weeks, and then stop ARVs for 56 weeks.

Participants in both study arms will restart ARVs regardless of STI duration if their viral load is above 50,000 copies/ml, they progress to CDC category C disease, or their CD4 count falls below 350 cells/mm3 or declines more than 50% from the last on-treatment CD4 level.

Step 2 will last 80 weeks. For the first year, participants will have study visits every 1 to 4 weeks, depending on whether they are taking ARVs. During the second year, participants will have study visits every 8 weeks. Study visits will include a brief medical history, blood and pregnancy tests, and voluntary behavioral questionnaires.

ELIGIBILITY:
Note: Step 2, Arm 3 has been eliminated as of 12/13/04.

Inclusion Criteria for Step 1:

* Acute or early HIV infection as defined by the study
* Agrees to use acceptable methods of contraception
* Agrees to begin antiretroviral treatment regimen within 21 days of diagnosis and no more than 3 days after study entry

Exclusion Criteria for Step 1:

* Unwilling to follow random assignment in Step 2
* Abnormal laboratory result within 21 days prior to study entry, unless abnormality is considered part of acute HIV infection
* Have taken antiretroviral drugs other than for postexposure prophylaxis (PEP). Patients who have undergone up to 30 days of previous PEP treatment are not excluded.
* Pregnancy or breastfeeding
* Previous participation in an HIV vaccine trial
* Previous use of experimental therapeutic immunizations or cytokine infusions

Inclusion Criteria for Participants Enrolling Directly into Step 2:

* Viral load of less than 400 copies/ml
* Enrolled in the AIEDRP CORE01 study, with stored blood samples obtained within 21 days prior to starting treatment on CORE01
* Currently receiving antiretroviral treatment regimen, with no interruptions for more than 7 consecutive days since the beginning of treatment
* Antiretroviral treatment was started within 21 days after HIV diagnosis
* Agrees to use acceptable methods of contraception

Exclusion Criteria for Step 2:

* Unwilling to follow random assignment to study arms and follow scheduled treatment interruptions
* More than 52 weeks of ARV treatment since diagnosis of acute/early HIV infection prior to entering Step 2
* CD4 count less than 350 cells/mm3 within 28 days of entry into Step 2
* AIDS-defining illness
* Pregnant or breastfeeding
* Previous participation in an HIV vaccine trial
* Previous use of experimental therapeutic immunizations or cytokine infusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Difference in mean HIV viral load between arms | At Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rosenberg, MD, Study Chair — Massachusetts General Hospital; Don Smith, MB, ChB, MD, Study Chair — University of New South Wales, Australia

REFERENCES:
- [Background] Girard PM, Schneider V, Dehee A, Mariot P, Jacomet C, Delphin N, Damond F, Carcelain G, Autran B, Saimot AG, Nicolas JC, Rozenbaum W. Treatment interruption after one year of triple nucleoside analogue therapy for primary HIV infection. AIDS. 2001 Jan 26;15(2):275-7. doi: 10.1097/00002030-200101260-00020. No abstract available. PMID 11216939
- [Background] Kaufmann GR, Zaunders JJ, Cunningham P, Kelleher AD, Grey P, Smith D, Carr A, Cooper DA. Rapid restoration of CD4 T cell subsets in subjects receiving antiretroviral therapy during primary HIV-1 infection. AIDS. 2000 Dec 1;14(17):2643-51. doi: 10.1097/00002030-200012010-00003. PMID 11125882
- [Background] Malhotra U, Berrey MM, Huang Y, Markee J, Brown DJ, Ap S, Musey L, Schacker T, Corey L, McElrath MJ. Effect of combination antiretroviral therapy on T-cell immunity in acute human immunodeficiency virus type 1 infection. J Infect Dis. 2000 Jan;181(1):121-31. doi: 10.1086/315202. PMID 10608758
- [Background] Markowitz M, Jin X, Hurley A, Simon V, Ramratnam B, Louie M, Deschenes GR, Ramanathan M Jr, Barsoum S, Vanderhoeven J, He T, Chung C, Murray J, Perelson AS, Zhang L, Ho DD. Discontinuation of antiretroviral therapy commenced early during the course of human immunodeficiency virus type 1 infection, with or without adjunctive vaccination. J Infect Dis. 2002 Sep 1;186(5):634-43. doi: 10.1086/342559. Epub 2002 Aug 9. PMID 12195350
- [Background] Walensky RP, Goldie SJ, Sax PE, Weinstein MC, Paltiel AD, Kimmel AD, Seage GR 3rd, Losina E, Zhang H, Islam R, Freedberg KA. Treatment for primary HIV infection: projecting outcomes of immediate, interrupted, or delayed therapy. J Acquir Immune Defic Syndr. 2002 Sep 1;31(1):27-37. doi: 10.1097/00126334-200209010-00004. PMID 12352147
- See also: Click here for more information on AIEDRP CORE01 — http://clinicaltrials.gov/ct/show/NCT00086372